CLINICAL TRIAL: NCT01083056
Title: Observational Study On Retinal Structure And Function Before And After Epimacular Membrane Peeling
Brief Title: Observational Study - ILM Peeling
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, M. Dominik Fischer, PD Dr. med. M. Dominik Fischer, University Hospital Tuebingen
Other Study IDs: ILM Peeling
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Epimacular Gliosis; Macular Hole
Keywords: retina; gliosis; macula; membrane; ILM
MeSH Terms: conditions — Retinal Perforations; Gliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Epimacular Gliosis Without Macular Hole
- Epimacular Gliosis With Macular Hole

SUMMARY:
This observational study investigates the effects of epimacular membrane peeling on the structure and function of the retina.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Epimacular Gliosis
* Must be scheduled for ILM-peeling independently of study
* Must be older then 18 years of age

Exclusion Criteria:

* Visual acuity > 0,4 logMAR (< 20/50 EDTRS)
* Other ophthalmological disorder affecting visual acuity and/or visual field and/or retinal structure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients at the University Eye Hospital Tuebingen
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
BCVA | 6 months after ILM peeling

CONTACTS AND LOCATIONS:
Overall Officials: Florian Gekeler, MD, Principal Investigator — Centre for Ophthalmology, University Hospital Tuebingen
Locations (1):
- Centre for Ophthalmology, University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany